CLINICAL TRIAL: NCT06249646
Title: Contained Hepatic Vascular Injuries Following Liver Trauma: a Retrospective Monocentric Study and Review of the Literature
Brief Title: Contained Hepatic Vascular Injuries Following Liver Trauma
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Urgences01
Record Dates: First submitted 2024-01-23; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Injury; Liver Injury; Pseudoaneurysm
MeSH Terms: conditions — Aneurysm, False

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: For thirty years, a major shift in the management of liver trauma has been seen. Contained hepatic vascular injuries (CHVI), including pseudo aneurysms and arteriovenous fistula, are often feared due to their risk of secondary bleeding. Nonetheless, knowledge of CHVI is scarce and no guidelines on their management have been set. The investigators aimed to validate the risk factors of CHVI, identify associated morbidities, and establish a management protocol.

Study Design: A retrospective study on 318 liver trauma from a level 1 trauma center over the last 15 years, comparing the presence or not of CHVI. Univarious and multivarious analyses were performed. A comparison of the management of CHVI was also performed.

ELIGIBILITY:
Inclusion Criteria:

* presence of liver trauma
* age above 15 years old
* a full contrast abdominal CT

Exclusion Criteria: none

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Liver trauma was identified on post-injury imaging evaluation or operative exploration. Admission following the trauma could either be directly from the trauma location or be a transfer from another regional hospital. Upon admission, if the patient was stable or stabilized following intensive care management, a contrast full-body CT scan was performed. Non-operative management was the primary treatment when possible. If the patient was unstable, primary surgical management was required. Surgical management could include sole exploration, hemostatic techniques, hepatic packing, drainage, or hepatectomy. If the investigators performed a damage control laparotomy with perihepatic packing, a second surgery was performed for definitive treatment after 24-48 h. In such cases, a contrast full-body CT scan was performed after the surgery. If a CT scan was not performed in the first 24 hours, the patient was not included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Identification of a % of CHVI on the initial or the follow-up Chest-Thorax scans. | 6 months
  A junior and a senior radiologist reviewed all initial and follow-up CT scans, blinded from the diagnostic.
  Contained hepatic vascular injuries (CHVI) was defined as Hepatic Pseudoaneurysm (HPA) and/or arterio-venous fistula (AVF), under the American Association for Surgery of Trauma (AAST) organ injury scale (2018 revision) for liver trauma definition: a contained focal collection of vascular contrast which decreases in attenuation on delayed phase images on contrast-enhanced CT

SECONDARY OUTCOMES:
Investigate the management of CHVI following liver trauma. | 6 months
  size in millimeters of pseudoaneurym conducting to angio-embolization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No